CLINICAL TRIAL: NCT07080762
Title: Microbiological and Clinical Efficacy of Photodynamic Therapy in Combination With Non-surgical Periodontal Therapy: a Clinical Trial
Brief Title: Photodynamic Therapy in Non-surgical Periodontal Therapy
Acronym: aPDT-PD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universita di Verona (Other)
Responsible Party: Principal Investigator, Alessia Pardo, PhD, Universita di Verona
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4242CESC; Ethics Committee (Registry Identifier: Ethics Committee for Clinical Trials of the Provinces of Verona and Rovigo)
Record Dates: First submitted 2025-07-09; First posted 2025-07-23 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-07

CONDITIONS: Photodynamic Therapy (PDT); Periodontitis; Antimicrobial Photodynamic Therapy
Keywords: Photodynamic Therapy; periodontitis
MeSH Terms: conditions — Periodontitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental : antimicrobial photodynamic therapy (aPDT) after non-surgical therapy (Experimental): The test group received antimicrobial photodynamic therapy (aPDT) immediately after non-surgical treatment. A diode laser with a wavelength of 660 nm was used (Helbo® TheraLite Laser, Bredent, Germany). The photosensitizer (Helbo® Biofilm Marker), based on phenothiazine chloride and supplied in pre-packaged sterile syringes, was delivered into the periodontal pocket using a sterile syringe with a flat tip. The photosensitizer was left in situ for 60 seconds. Subsequently, all periodontal pocket walls were irradiated for ten seconds each (disto-lingual, lingual, mesio-lingual, mesio-buccal, buccal, disto-buccal), for a total duration of 60 seconds.
  Interventions: Device: antimicrobial photodynamic therapy (aPDT) after non-surgical therapy
- No intervention: non-surgical therapy (No Intervention): In the control group, non-surgical periodontal therapy was performed using both mechanical and manual instrumentation with curettes and ultrasonic devices.

INTERVENTIONS:
Device: antimicrobial photodynamic therapy (aPDT) after non-surgical therapy — In the test, a photoactive substance activated with laser light (20 mW, 660 nm) was applied to the post-non-surgical site for 60 seconds to promote disinfection Other Name: antimicrobial photodynamic therapy (aPDT) after non surgical therapy
  Arms: Experimental : antimicrobial photodynamic therapy (aPDT) after non-surgical therapy

SUMMARY:
Non-surgical periodontal therapy is a widely adopted procedure for the treatment of periodontitis, particularly in its moderate to severe stages. The approach involves the mechanical and manual debridement of subgingival biofilm and calculus through the use of ultrasonic scalers and hand curettes. This method aims to disrupt the pathogenic bacterial load within periodontal pockets and promote clinical attachment gain while reducing inflammation. However, the mechanical removal of biofilm alone may not always ensure complete bacterial eradication, especially in deep or anatomically complex sites.

To enhance bacterial disinfection and optimize clinical outcomes, adjunctive use of antimicrobial photodynamic therapy (aPDT) has been introduced. aPDT is a non-invasive technique that involves the activation of a photosensitizing agent by light at a specific wavelength, leading to the production of reactive oxygen species capable of selectively damaging microbial cells. This reaction occurs without affecting surrounding healthy tissues and has been shown to be effective against a broad spectrum of periodontal pathogens.

The synergistic effect of combining conventional non-surgical periodontal therapy with aPDT allows for a more comprehensive decontamination of periodontal pockets. In particular, aPDT contributes to the disruption of residual bacterial biofilm that may persist after mechanical instrumentation, thereby potentially improving both short- and long-term periodontal stability. In addition to its antimicrobial action, aPDT may exert a biostimulatory effect, enhancing tissue healing through increased local microcirculation and cellular activity.

This study aims to evaluate the clinical efficacy of adjunctive antimicrobial photodynamic therapy following non-surgical periodontal treatment in patients with severe periodontitis. The protocol involves initial subgingival instrumentation using ultrasonic and manual tools, followed by the application of a photosensitizer and subsequent laser activation within the periodontal pockets. The hypothesis of this study is that the addition of aPDT provides superior bacterial reduction and improved clinical outcomes compared to mechanical therapy alone.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 84 years;
* Good general health status;
* Diagnosis of severe periodontitis involving at least 30% of all teeth, with at least three non-adjacent teeth presenting three sites with probing pocket depth (PPD) greater than 4 mm in at least two quadrants, and having lost at least four teeth due to periodontitis;
* Presence of at least 16 teeth, with a minimum of four teeth per quadrant.

Exclusion Criteria:

* Pregnancy or breastfeeding;
* Presence of decompensated systemic diseases that may compromise the outcomes of the study or the patient's health;
* Regular use of antibiotics;
* Regular use of anti-inflammatory drugs (NSAIDs, corticosteroids, or aspirin);
* Use of anticoagulant medications;
* History of systemic antibiotic therapy within six months prior to enrollment;
* History of any periodontal therapy within six months prior to enrollment;
* Presence of severe mental or cognitive disorders.

Ages: 18 Years to 84 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2023-11-03 (Actual); Primary Completion 2024-05-30 (Actual); Study Completion 2024-05-30 (Actual)

PRIMARY OUTCOMES:
Probing Pocket Depth PPD Index | T0 (Baseline), T1(7 days after baseline), T2 (14 days after baseline), T3 (3 months after baseline)
  Probing depth is the distance from the gingival margin to the base of the pocket (mm)
Microbiological analysis | T0 (Baseline), T2 (14 days after baseline), T3 (3 months after baseline)
  The microbiological analysis qualitatively (yes/no) assesses the presence of six types of periodontopathogenic bacteria (Aggregatibacter actinomycetemcomitans, Porphyromonas gingivalis, Prevotella intermedia, Tannerella forsythia, Treponema denticola, Actinomyces naeslundii) using sterile paper points inserted into the periodontal pocket prior to non-surgical periodontal therapy. For each site analyzed, two saliva samples are collected: one is placed in a test tube containing ethanol, and the other in a tube containing ammonium thioglycolate. The samples are subsequently transported to the microbiology department of the Integrated University Hospital of Verona for analysis.

SECONDARY OUTCOMES:
Recession REC Index | T0 (Baseline), T1(7 days after baseline), T2 (14 days after baseline), T3 (3 months after baseline)
  Recession is the apical shift of the marginal tissues associated with the attachment loss exposing the root or implant surface to the oral environment (mm)
Clinical attachment level CAL Index | T0 (Baseline), T1(7 days after baseline), T2 (14 days after baseline), T3 (3 months after baseline)
  measured in mm as distance from the CEJ to the gingival margin (GM)
Plaque Index | T0 (Baseline), T1(7 days after baseline), T2 (14 days after baseline), T3 (3 months after baseline)
  This index ascertains the thickness of plaque along the gingival margin (%)
Bleeding on probing BOP Index | T0 (Baseline), T1(7 days after baseline), T2 (14 days after baseline), T3 (3 months after baseline)
  is an indicator of tissue inflammatory response to bacterial pathogens (%)

CONTACTS AND LOCATIONS:
Locations (1):
- Alessia Verona, Verona, VR, Italy